CLINICAL TRIAL: NCT06496698
Title: Impact of Suture Technique on Wound Healing in Ankle Fracture Surgery: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117966
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcuticular Suture Group (Experimental): Running subcuticular Vicryl 3-0 sutures will be placed on patients in the experimental group.
  Interventions: Procedure: Subcuticular Suture
- Simple Interrupted Suture Group (Active Comparator): Simple interrupted Monocryl 3-0 sutures will be placed on patients in the control group.
  Interventions: Procedure: Simple Interrupted Suture

INTERVENTIONS:
Procedure: Simple Interrupted Suture — In the control group, simple interrupted sutures will be used for wound closure after surgical repair of ankle fractures.
  Arms: Simple Interrupted Suture Group
Procedure: Subcuticular Suture — In the experimental group, subcuticular sutures will be used for wound closure after surgical repair of ankle fractures.
  Arms: Subcuticular Suture Group

SUMMARY:
Our primary aim is to compare the complication rates of patients with ankle fractures who underwent skin closure using a running subcuticular suture pattern compared to an interrupted suture pattern. At the time of the operation, participants will be assigned to either the Subcuticular Suture Group (SSG) or the Simple Interrupted Suture Group (SISG) using computer-generated randomization programs. The surgeon will perform the assigned closure technique using standardized techniques. Running subcuticular Vicryl 3-0 sutures will be placed on patients in the experimental group while simple interrupted Monocryl 3-0 sutures patients in our control group.

Patients will be followed up at the two-week and eight-week postoperative mark where we will use the Patient and Observer Scar Assessment Scale (POSAS) to evaluate and compare wound healing. Additionally, photographs of the scars will be captured to visually assess the healing progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or older with isolated ankle fractures requiring surgical intervention and who consent to participate.

Exclusion Criteria:

* Patients that will be excluded from this study include those with complex ankle fractures, open fractures, a history of wound healing disorders, and/or those unable to provide consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication rates | 2 and 8 weeks post-op.
  Complications include wound infection, dehiscence, suture breakage, suture abscess, necrosis, allergic reactions, malunion, hardware failure, and the need for reoperation or revision surgery.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | 2 and 8 weeks post-op.
  The Patient and Observer Scar Assessment Scale (POSAS) is a comprehensive tool used to evaluate the quality of scars from both the patient's and observer's perspectives. It consists of two parts: the Patient Scale and the Observer Scale.
Self-reported foot and ankle score (SEFAS) | 2 and 8 weeks post-op.
  Consists of 12 items related to pain, limping, swelling, and use of orthotics and walking.

IPD SHARING:
Plan to Share IPD: Undecided